CLINICAL TRIAL: NCT07181863
Title: Bridging Gaps, Enhancing Wellbeing: Examining the Effectiveness of the Technology-Enabled Collaborative Care for Diabetes and Mental Health (TECC-DM) Model
Brief Title: Technology-Enabled Collaborative Care for Diabetes and Mental Health
Acronym: TECC-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Centre for Addiction and Mental Health (Other); Diabetes Canada (Other)
Responsible Party: Principal Investigator, Carly Whitmore, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19043
Record Dates: First submitted 2025-09-08; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Mental Health; Diabetes Distress
Keywords: type 2 diabetes; diabetes distress; technology; collaborative care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: TECC-DM is a relation-driven, integrated care model delivered through accessible technology (phone, text, Zoom, REDCap). Participants in the experimental group (n=80) meet weekly with a health coach, who supports motivation, goal-setting, behaviour change, and care navigation without providing direct pharmacological care. Coaches identify mental health needs, liaise with an interdisciplinary virtual care team, and map services and referrals. Weekly ~1-hour sessions focus on building therapeutic relationships, prioritizing behaviour change, and enhancing self-management. A virtual care team, comprised of interprofessional healthcare team members, meets with the coach to provide guidance. TECC-DM complements but does not replace usual diabetes care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECC-DM model (Experimental): Participants (n=80) are randomized to the TECC-DM arm, a 12-week, relation-driven and integrated model of care delivered virtually in addition to usual diabetes care. Weekly 1-hour sessions with a health coach are supported by guidance from an interdisciplinary virtual care team, using phone, text, Zoom, and REDCap. The program follows a structured protocol to ensure fidelity. TECC-DM is designed to improve quality of life (primary outcome) and goals of care (secondary outcomes: mental health, self-management, and physiological indicators).
  Interventions: Behavioral: Health coaching
- Educational emails (Active Comparator): Participants (n=80) receive usual diabetes care, which may include primary or specialist care and community-based supports, with services documented to capture variation. In addition, participants receive 10 standardized educational emails over 12 weeks. This arm provides a structured, fidelity-monitored comparison to TECC-DM.
  Interventions: Other: Educational emails

INTERVENTIONS:
Behavioral: Health coaching — Health coaching is the active component of TECC-DM. In weekly 1-hour sessions, the coach builds a therapeutic relationship, supports goal-setting and behaviour change, addresses mental health needs, coordinates resources, and empowers participants to navigate care. Coaching is delivered according to a standardized protocol, in consultation with the virtual care team, and targets improvements in quality of life and goals of care. Coaches do not provide pharmacological treatment or replace usual diabetes care.
  Arms: TECC-DM model
Other: Educational emails — Participants receive usual diabetes care (e.g., primary care, endocrinology, community supports) plus 10 standardized educational emails over 12 weeks, delivered according to a consistent protocol. Unlike TECC-DM, this approach does not involve a therapeutic relationship, health coach, or interdisciplinary care team.
  Arms: Educational emails

SUMMARY:
Managing both type 2 diabetes and mental health challenges can be difficult, and many people do not receive care that supports both. This study looks at how virtual health coaching and support from interdisciplinary care teams can help people better manage their health.

The purpose of this study is to test the effectiveness of a virtual health coaching program for adults living with type 2 diabetes and mental health challenges compared to usual care. The Technology-Enabled Collaborative Care for type 2 Diabetes and Mental health (TECC-DM) program includes weekly coaching calls, support from an interdisciplinary care team, and online tools to aid self-management. The findings from this study will be used to help improve services for people who have type 2 diabetes and co-occurring mental health symptoms.

DETAILED DESCRIPTION:
This research will:

Implement and evaluate a relation-driven care solution that integrates physical and mental healthcare for adults living with type 2 diabetes (T2D) and comorbid mental health challenges. Applying the principles of relation-centred care which expands patient-centred care to all team members involved, the TECC-DM model was co-designed to improve collaborative care between and across sectors, settings, and professionals. This model enhances the core relationship between provider and patients while empowering the person to be an active agent in their health and care.

Assess the effectiveness of the TECC-DM intervention (n=80) on patient-relevant (quality of life) and provider-level (satisfaction) outcomes compared to usual care (n=80). Drawing upon established feasibility data, and delivered in addition to existing diabetes care, the TECC-DM model of care may address important health system challenges in primary care, including those related to access, resources, and skill mix, while delivering whole-person care.

Study the implementation of the TECC-DM model alongside its effectiveness. Engaging a partner advisory group, knowledge users, and clinicians reflects the shared values of our team and ensures that this research leverages a wealth of expertise and real-world insights to inform future applications.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Diagnosed with type 2 diabetes (T2D)
* Experiencing mental health challenges, defined as:
* Hospital Anxiety and Depression Scale (HADS) score ≥8 on either subscale OR
* Diabetes Distress Scale (DDS) score ≥2
* Community-living
* Able to communicate verbally in English
* Residing in Ontario during study participation

Exclusion Criteria:

* Diagnosis of severe mental illness (e.g., schizophrenia, psychotic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | From baseline to 12 weeks post-intervention and at 6-month follow-up
  Quality of life refers to an individual's overall well-being, encompassing physical, mental, emotional, and social dimensions of health. In this study, it is measured using the EuroQol-5D (EQ-5D), which captures participants' perceptions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Unit of Measure: EQ-5D-5L index score. Minimum Value: 0 (the worst possible health state). Maximum Value: 100 (the best possible health state). Interpretation: Higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Change in diabetes distress score (Diabetes Distress Scale, DDS) | From baseline to 12 weeks post-intervention and at 6-month follow-up
  The DDS measures the emotional burden, regimen distress, interpersonal distress, and physician distress related to living with diabetes. Scores range from 1-6, with higher scores indicating greater distress. Outcome will be reported as mean change in total and subscale scores from baseline to 12 weeks and 6 months, with the proportion of participants achieving a clinically meaningful reduction (≥0.5 points) also reported.
Change in psychological and behavioural health symptoms (Global Appraisal of Individual Needs Short Screener, GAIN-SS) | From baseline to 12 weeks post-intervention and at 6-month follow-up
  The GAIN-SS is a validated screener for internalizing and externalizing disorders, substance use, and crime/violence problems. Scores range from 0-15 per subscale, with higher scores indicating more symptoms. Outcome will be reported as change in total and domain scores from baseline to 12 weeks and 6 months, along with the number of participants with reduced symptom severity.
Change in perceived stress score (Perceived Stress Scale, PSS) | From baseline to 12 weeks post-intervention and at 6-month follow-up
  The PSS measures the degree to which situations in one's life are appraised as stressful, with scores ranging from 0-40. Higher scores indicate greater perceived stress. Outcome will be reported as change in mean score from baseline to 12 weeks and 6 months, with distribution of participants across mild, moderate, and high stress categories also described.
Change in depressive symptoms (Patient Health Questionnaire, PHQ-9) | From baseline to 12 weeks post-intervention and at 6-month follow-up
  The PHQ-9 measures the presence and severity of depressive symptoms, with scores ranging from 0-27. Higher scores indicate more severe depression. Outcome will be reported as change in mean score from baseline to 12 weeks and 6 months, and the proportion of participants achieving clinically significant improvement (≥5-point reduction or remission, score <5).
Change in diabetes self-management (Diabetes Self-Management Questionnaire, DSMQ) | From baseline to 12 weeks post-intervention and at 6-month follow-up
  The DSMQ assesses key self-management domains including glucose monitoring, medication adherence, diet, and physical activity. Scores range from 0-10, with higher scores indicating more effective self-management. Outcome will be reported as change in total and subscale scores from baseline to 12 weeks and 6 months.
Change in technology-enabled self-management behaviour (Diabetes Self-Management Technology Questionnaire) | From baseline to 12 weeks post-intervention and at 6-month follow-up
  This questionnaire assesses use and integration of diabetes technologies such as continuous glucose monitoring, insulin pumps, and mobile applications. Higher scores indicate more frequent or effective use of technology for self-management. Outcome will be reported as change in mean scores from baseline to 12 weeks and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Carly Whitmore, RN PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of health and mental health information, the risk of re-identification, and ethical requirements under local privacy legislation and research ethics board approvals. Aggregated data may be available upon reasonable request.

REFERENCES:
- [Background] Vojtila L, Sherifali D, Dragonetti R, Ashfaq I, Veldhuizen S, Naeem F, Agarwal SM, Melamed OC, Crawford A, Gerretsen P, Hahn M, Hill S, Kidd S, Mulsant B, Serhal E, Tackaberry-Giddens L, Whitmore C, Marttila J, Tang F, Ramdass S, Lourido G, Sockalingam S, Selby P. Technology-Enabled Collaborative Care for Concurrent Diabetes and Distress Management During the COVID-19 Pandemic: Protocol for a Mixed Methods Feasibility Study. JMIR Res Protoc. 2023 Jan 17;12:e39724. doi: 10.2196/39724. PMID 36649068
- [Background] Sherifali D, Whitmore C, Naeem F, Melamed OC, Dragonetti R, Kouzoukas E, Marttila J, Tang F, Tanzini E, Ramdass S, Selby P. Technology-Enabled Collaborative Care for Type-2 Diabetes and Mental Health (TECC-D): Findings From a Mixed Methods Feasibility Trial of a Responsive Co-Designed Virtual Health Coaching Intervention. Int J Integr Care. 2024 Feb 16;24(1):12. doi: 10.5334/ijic.7608. eCollection 2024 Jan-Mar. PMID 38370569